CLINICAL TRIAL: NCT04068909
Title: Exacerbation of Coronary Heart Disease: the Logic and Probabilistic Processes of Flow Prediction for Optimization of Treatment
Brief Title: ObseRvation After Acute Coronary Syndrome for deveLopment of trEatment Options
Acronym: ORACLE
Status: Completed | Type: Observational
Sponsor: Central State Medical Academy (Other)
Responsible Party: Principal Investigator, Larisa Minushkina, professor, Central State Medical Academy
Other Study IDs: ORACLE-II
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2019-08

CONDITIONS: Acute Coronary Syndrome
Keywords: coronary artery disease; death; gene; bleeding; atherosclerosis
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Death; Hemorrhage; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples for DNA analysis in ethylenediaminetetraacetic acid (EDTA)vacutainer tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute coronary syndrome: All patients should receive standard therapy for acute coronary syndrome and concomitant diseases. All drugs are prescribed according current guidelines and approved indications.

SUMMARY:
The aim of the study is developing an individualized risk model for the unfavorable outcomes of coronary artery disease and complications from ongoing therapy, according to clinical, instrumental, biochemical and genetic parameters in patients with acute coronary syndrome.

Inclusion criteria: patients with acute coronary syndrome (with or without ST elevation) who have indications for PCI Number of inclusion patients - 1655 patients Scheduled time of follow up - 24 month Primary end-point: all-cause death Secondary end-points: any cardiovascular events (cardiovascular death, nonfatal myocardial infarction, non-fatal stroke); non-fatal myocardial infarction; recurrent acute coronary syndrome; non-fatal stoke; complicated atherosclerosis; recurrent PCI; bleeding

DETAILED DESCRIPTION:
The role of genetic factors in the development of coranary heart disease (CHD) exacerbations studied not enough. Most research in this area planned and carried out on a "case-control". Using a similar protocol entails significant errors are associated with a high incidence of subclinical atherosclerotic vascular lesions. Moreover, much of atheroma is extravasal, making it impossible to identify them by angiography. Therefore, necessary to conduct prospective studies to estimate the frequency of so-called hard endpoints. Previously, similar trials were conducted, mainly in connect with drug approving procedures. The spread data from them to other patients directly is not entirely justified. At the same time, the influence of genetic factors in this group of patients can be substantial.

In the previous part of the study, the sample of patients of Moscow, St. Petersburg, Kazan, Chelyabinsk, Stavropol, Perm, and Rostov-on-the-Don was formed, of 1,200 people admitted due to acute coronary syndrome (ACS) including unstable angina and acute myocardial infarction, at coronary care units with follow-up for three years. We found several factors, including genetic, that significantly affect the outcomes of the disease. Coronary atherosclerosis and its complications now considered as a multifactorial disease associated with inherent factors. Therefore, the project provides, besides accounting a significant amount of clinical and instrumental data, the determination of a wide range of genotypes and alleles of polymorphic markers candidate genes encoding the protein factors of the hemostatic system, enzymes of lipid metabolism system, and anti-inflammatory cytokines. It is assumed that the prediction outcomes of coronary heart disease should be carried out taking into account the fact that several factors (gender, diabetes, age, aortic stenosis, atrial fibrillation, etc.) can not only significantly change the forecast itself but also affecting the significance of other risk factors. Since the last study, the standards significantly of ACS management changed. Invasive treatment not only creates opportunities to reduce coronary mortality but also increased demands on the patient's adherence to the assigned medication and creates additional risks associated with its activity (especially with an antithrombotic treatment activity). In these circumstances, the development of personalized approaches to prescribing drugs is particularly important. Thus, the prediction of coronary heart disease outcomes after an ACS on a set of clinical, instrumental, biochemical and genetic indicators is of great importance, as it allows to plan the most optimal treatment for the individual patient.

The aim of the study was to develop a model of individualized risk of coronary heart disease outcomes and side effects of therapy based on clinical and instrumental, biochemical, and genetic parameters in patients with ACS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute coronary syndrome without ST-segment elevation meeting the criteria of a very high, high or intermediate risk, and patients from the low-risk group, if they have episodes of myocardial ischemia in any way Very high risk (1 criterion is sufficient)

   * Pulmonary edema, most probably due to ischemia.
   * The newly appears or increased noise of mitral regurgitation.
   * Rhythm of the gallop, newly developed or intensified wheezing in the lungs.
   * Hypotension against ischemia
   * Ischemia refractory to treatment
   * Persistent ventricular tachycardia or the occurrence of ventricular rhythm disturbances during an attack of ischemia High risk

     (1 criterion is sufficient)
   * An anginal attack more than 20 minutes within the next 48 hours before admission
   * Transitional elevations ST (duration less than 20 min)
   * GRACE score > 140 points
   * Increased cardiospecific markers of necrosis. (you must have at least 2 criteria)
   * Age> 75 years.
   * Angina pectoris with transient changes ST> 0.05 mV.

   Intermediate risk (1 criterion is sufficient)
   * Age> 75 years.
   * Angina pectoris with transient changes ST> 0.05 mV.
   * Inversion of the T wave on ECG (≥ 0.2 mV).
   * GRACE score 104-139 points

   (it is necessary to have at least 2 criteria)
   * Angina of rest (<20 min), stopped spontaneously or with the help of nitroglycerin (NG).
   * Anamnesis of pathology of peripheral or cerebral arteries,
   * Postponed myocardial infarction, including painless, history of revascularization (PCI or CABG)
   * Diabetes.
   * Chronic renal failure (GFR <50 mL / min)

   Low risk All other patients with suspicion of ACS require a survey to identify episodes of ischemia
2. Patients with acute coronary syndrome with ST-segment elevation

   Patients who were hospitalized with symptoms due to acute myocardial infarction (the duration of infarction is no more than 10 days, by the time of hospitalization) and at least one of the following additional criteria identified upon admission to hospital:
   * ST elevation: a persistent ST increase of 1 mm in two adjacent leads from the limbs, or an ST increase of 2 mm in two adjacent thoracic leads
   * the appearance of a new left bundle branch block
   * dynamics of acute myocardial infarction
3. Signed informed consent to participate in the study

Exclusion Criteria:

* Lack of patient consent to participate in the study
* Impossibility of contact with the patient after discharge after index event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of consistently hospitalized patients with ACS from 4 vascular centers of Moscow, Kazan, Astrakhan and Krasnodar
Sampling Method: Probability Sample
Enrollment: 1655 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
all-cause death | Number of Participants with end-point during 360 days
  death from any cause

SECONDARY OUTCOMES:
cardiovascular events | Number of Participants with end-point during 360 days
  cardiovascular death, non-fatal myocardial infarction, non-fatal stroke
non-fatal myocardial infarction | Number of Participants with end-point during 360 days
  non-fatal myocardial infarction
recurrent acute coronary syndrome | Number of Participants with end-point during 360 days
  all cases of recurrent myocardial infarction or unstable angina after the index events
recurrent PCI | Number of Participants with end-point during 360 days
  all cases of recurrent PCI after the index hospitalization
complicated atherosclerosis | Number of Participants with end-point during 360 days
  peripheral atherosclerosis need hospitalisation
non-fatal stroke | Number of Participants with end-point during 360 days
  all cases of non-fatal stroke

OTHER OUTCOMES:
bleeding | Number of Participants with end-point during 360 days
  all cases of bleeding during and after the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry A Zateyshchikov, prof, Principal Investigator — Central State Medical Academy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brazhnik VA, Minushkina LO, Boeva OI, Khasanov NR, Kosmacheva ED, Chichkova MA, Zateyshchikov DA. Risk Stratification after an Acute Coronary Syndrome: Significance of Antithrombotic Therapy. J Clin Med. 2021 Apr 8;10(8):1572. doi: 10.3390/jcm10081572. PMID 33917922

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04068909/Prot_SAP_000.pdf